CLINICAL TRIAL: NCT06599554
Title: Outcome And Complications Assessment In The Surgical Treatment Of Distal Fibular Fractures: an Observational Study
Brief Title: Outcome And Complications Assessment In The Surgical Treatment Of Distal Fibular Fractures
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Principal investigator, Istituto Ortopedico Rizzoli
Other Study IDs: ANKLE-FRACT
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Ankle Fractures
Keywords: ankle injuries; ankle fractures; foot surgery
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: patients suffering from fibula fracture treated surgically through reduction and synthesis with an anatomical fibula plate
  Interventions: Other: follow up scores

INTERVENTIONS:
Other: follow up scores — The radiological reports will be read, analyzing when the bony consolidation of the fracture is reported in relation to the time elapsed since the operation.
  The questionnaires will be submitted to all patients who have completed the course at 1 year.
  All patients who sign the informed consent will be asked to complete the questionnaires either at the time of the follow-up visit by common clinical practice or by telephone, in the event that the patients have exceeded the 1-year follow-up

SUMMARY:
From the archives of the IRCCS Rizzoli Orthopedic Institute (SIR2020) all cases of patients undergoing surgical interventions for the reduction and synthesis of fractures of the distal fibula will be retrieved Ankle-fract Version 2.0 8/08/2024 7 isolated or associated with other lesions, treated surgically with placement of anatomical fibula plates and any accessory procedures from 01/01/2019 to 1/1/2024. An overall electronic database will be created and all medical records of these cases will be reviewed.

The pre- and post-operative data of the patients will be analyzed by analyzing the medical records and the post-operative x-rays (x-ray performed as per common clinical practice, present at the institute (IRCCS Istituto Ortopedico Rizzoli) which highlight consolidation of the fracture.

The radiological reports will be read, analyzing when the bony consolidation of the fracture is reported in relation to the time elapsed since the operation.

The questionnaires will be submitted to all patients who have completed the course at 1 year.

All patients who sign the informed consent will be asked to complete the questionnaires either at the time of the follow-up visit by common clinical practice or by telephone, in the event that the patients have exceeded the 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from fibula fracture treated surgically through reduction and synthesis with an anatomical fibula plate;

  * patients of both sexes aged between 18-90 years;
  * patients who have given their written informed consent to participate in the study Patients in possession of a post-operative control x-ray examination to evaluate consolidation and alignment (x-ray performed as per common clinical practice).

Exclusion Criteria:

* patients with severe postural instability;

  * Patients incapable of understanding or wanting;
  * patients with concomitant neurological pathologies that prevent walking and standing
  * bedridden patients.
  * Lack of written informed consent to participate in the study
  * written form to participate in the study
  * Physiotherapy not performed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery for reduction and synthesis of fibula fracture treated with anatomical fibula plate from 01/01/2019 to 01/01/2024 operated at SC Orthopedic and Traumatology Clinic II, with minimum follow-up of 1 year, with possibly associated with other surgical procedures made necessary due to the trauma
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Disability Index | after 1 year
  It is a self-reported questionnaire used to assess functional limitations and disabilities associated with foot and ankle conditions. The FADI consists of two parts: the main part with 26 questions and the additional sports module with 8 questions. Each question is rated on a 5-point scale (0 to 4), with 0 indicating the most difficulty and 4 indicating no difficulty. The scores for each question are added and converted to a percentage, with a higher percentage indicating better function. It is rated on a total of 104 points, with a score of 0 indicating maximum disability and a score of 104 indicating no disability

SECONDARY OUTCOMES:
The American Orthopedic Foot and Ankle Score | after 1 year
  clinical and functional evaluation for ankle and foot most validated and used in literature. There are 4 versions depending on the anatomical region to be evaluated: ankle and hindfoot, midfoot, first toe, last 4 toes. In this case the ankle and hindfoot version will be used. The score consists of 9 questions grouped into 3 categories for a total of 100 maximum points: Pain (up to 40 points), Function (up to 50 points) and Alignment (up to 10 points); 100 points represent the best possible clinical-functional condition and the absence of symptoms, 0 points represent the worst possible clinical-functional condition. It is a tool that combines the subjective component of the patient with the objective evaluation by the doctor.
Visual Analog Score | after 1 year
  visual representation of the extent of pain that the patient subjectively feels. The VAS is represented by a 10 cm long line in the original validated version, with or without notches corresponding to each centimeter. One end indicates the absence of pain and corresponds to 0, the other end indicates the worst pain imaginable and corresponds to 10. The scale is filled in manually by the patient who is asked to draw a sign on the line that represents the perceived pain . The distance measured from the 0 end corresponds to the subjective measurement of pain.
12-Item Short Form Survey | after 1 year
  short version of the SF-36 questionnaire (link). Through 12 of the 36 questions of the original questionnaire it allows us to investigate the two synthetic indices, PCS Physical Component Summary for the Physical State and MCS Mental Component Summary for the Mental State. The greatest strengths of this questionnaire are its brevity and relative ease of use. In Italy the questionnaire was used among other things in 2000 in a multipurpose ISTAT survey on the health status of Italians and a reference database is available with data on a sample of 61,434 subjects representative of the Italian population. Even for this short form, the literature is full of experiences and studies that demonstrate its validity and reliability.
EQ-5D (EuroQoL) Current Health Assessment | after 1 year
  valid tool for measuring a patient's quality of life.
x-rays analysis | after 1 year
  the radiological reports will be read, analyzing when the bony consolidation of the fracture is reported in relation to the time elapsed since the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided